CLINICAL TRIAL: NCT04772976
Title: The Relationship Between Dietary Phytochemical Index, Oxidative Stress and Inflammation of Patients With Ankylosing Spondylitis
Brief Title: Relationship Between Diet, Oxidative Stress and Inflammation in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatma Gül Yurdakul, Associate Professor, Ankara City Hospital Bilkent
Other Study IDs: E1-20-938
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Antioxidant capacity; Diet; Phytochemical index; Oxidant capacity
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Patients with Ankylosing Spondylitis
  Interventions: Other: Observational study, not applicable
- Healthy controls: Healthy controls
  Interventions: Other: Observational study, not applicable

INTERVENTIONS:
Other: Observational study, not applicable — Observational study, not applicable

SUMMARY:
Ankylosing Spondylitis (AS) is a chronic inflammatory autoimmune disease. The aim of this study is to reveal the relationship between dietary intake, blood total antioxidant capacity and disease activity in individuals with AS. This study will include patients diagnosed with AS who applied to Ankara City Hospital Physical Therapy and Rehabilitation Hospital, and a control group that does not have AS. The sociodemographic characteristics and nutritional habits and 1-day physical activity status of individuals with AS and healthy persons will be recorded. Anthropometric measurements of all individuals (such as height length (cm) and body weight) will be taken. From the height and body weight measurements, the individuals body mass indexes will be calculated. All parts of the questionnaire for individuals included in the research will be filled in by the researcher through face-to-face interview technique. The disease activity score of the individuals in the case group will be evaluated by the physician. Serum biochemical parameters will be taken from the patient files. In the patient information system of the control group, above mentioned blood tests will be recorded from the examinations performed in the last 1 month. Serum total antioxidant and oxidant levels will be measured in a private laboratory with a tube (5 ml) of blood from all individuals. The parameters to be examined in blood samples are specific to the study and their cost will be covered by the researchers.

DETAILED DESCRIPTION:
Ankylosing Spondylitis (AS) is a chronic inflammatory autoimmune disease that progresses with inflammation of synovial membranes. The aim of this study is to reveal the relationship between total dietary phytochemical intake, blood total antioxidant capacity and disease activity in individuals with AS. This study will include patients diagnosed with AS who applied to Ankara City Hospital Physical Medicine and Rehabilitation Hospital, and a control group that does not have AS and that meet exclusion criteria. The sociodemographic characteristics and nutritional habits, one-day food consumption records and 1-day physical activity status of AS diagnosed and healthy individuals included in the study will be recorded with a questionnaire. Anthropometric measurements of all individuals (case and control) such as height length (cm) and body weight (kg) will be taken. From the height and body weight measurements, the students' body mass indexes will be calculated from the formula [weight (kg) / height (m²)]. Waist circumference; The perimeter passing through the middle of the distance between the lowest costa and crista iliaca superior will be measured by tape measure. All parts of the questionnaire for individuals included in the research will be filled in by the researcher through face-to-face interview technique. The disease activity score (ASDAS) of the individuals in the case group will be evaluated by the physician. Serum biochemical parameters (complete blood count, fasting blood sugar, liver function tests, urea, creatinine, lipid profile, erythrocyte sedimentation rate, c-reactive protein) will be taken from the patient files. In the patient information system of the control group, complete blood count, fasting blood sugar, liver function tests, urea, creatinine, lipid profile, erythrocyte sedimentation rate, and c-reactive protein levels will be recorded from the examinations performed in the last 1 month. Serum total antioxidant and oxidant levels will be measured in a private laboratory with a tube (5 ml) of blood from all individuals. After the blood samples are centrifuged, 0.5 ml will be separated into eppendorfs. Samples will be stored in a -80 degree refrigerator in the Physical Medicine and Rehabilitation Hospital. Total antioxidant and oxidant capacity measurement will be done in a private laboratory in Ankara in the form of service procurement by Erel method. Samples for total antioxidant and oxidant analysis will be sent to the relevant laboratories in dry ice. The parameters to be examined in blood samples are specific to the study and their cost will be covered by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being followed up with a diagnosis of AS

Exclusion Criteria:

* Individuals under 18 and over 65 years of age,
* Those with active or previous history of malignancy
* Those diagnosed with cardiovascular disease
* Those with chronic kidney disease
* Those with liver disease
* Those with acute or chronic inflammatory diseases
* Those with diabetes
* Those with acute or chronic infections
* Those who consume alcohol,
* Smokers,
* Pregnant and breastfeeding women,
* People with severe psychiatric illness,
* Those who take regular medication and antioxidant nutritional supplements,
* Those who are not volunteer to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic patients
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Dietary phytochemical index | Will be done only once on the first day after inclusion.
  Dietary phytochemical index is calculated from one day dietary record. Higher index is better.
Total antioxidant and oxidant capacity | Blood samples will be obtained once on the first day after inclusion. Samples will be stored in -80 C medical refrigerator and analysis will be done after collection of all samples.
  Higher total antioxidant capacity and lower oxidant capacity is better.
Ankylosing Spondylitis Disease Activity Score | Will be done only once on the first day after inclusion.
  Higher scores (>2.1) mean active disease. Lower scores (<1.3) mean inactive disease

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gul Yurdakul, Assoc.Prof., Principal Investigator — Ankara City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara, Turkey; Hatice Bodur, Prof., Principal Investigator — Ankara City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara, Turkey; Evren Yasar, Prof, Principal Investigator — Ankara City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara, Turkey; Nilgun Seremet Kurklu, Asist.Prof., Principal Investigator — Akdeniz University, Faculty of Health Sciences, Department of Nutrition and Dietetics; Kubra Tel Adiguzel, Asist.Prof., Principal Investigator — University of Health Sciences Turkey, Gulhane Faculty of Health Sciences, Nutrition and Dietetics
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feijoo M, Tunez I, Tasset I, Montilla P, Ruiz A, Collantes E. Infliximab reduces oxidative stress in ankylosing spondylitis. Clin Exp Rheumatol. 2009 Jan-Feb;27(1):167-8; author reply 168. No abstract available. PMID 19327250
- [Background] Karakoc M, Altindag O, Keles H, Soran N, Selek S. Serum oxidative-antioxidative status in patients with ankylosing spondilitis. Rheumatol Int. 2007 Oct;27(12):1131-4. doi: 10.1007/s00296-007-0352-3. Epub 2007 Apr 19. PMID 17443328
- [Background] Howes MJ, Simmonds MS. The role of phytochemicals as micronutrients in health and disease. Curr Opin Clin Nutr Metab Care. 2014 Nov;17(6):558-66. doi: 10.1097/MCO.0000000000000115. PMID 25252018